CLINICAL TRIAL: NCT04571281
Title: Dynamics of the Capillary Lactate Levels in Patients With Out-of-hospital Cardiac Arrest
Brief Title: Dynamics of the Capillary Lactate Levels in OHCA
Status: Completed | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Matej Strnad, Assoc. Professor, University Medical Centre Maribor
Other Study IDs: KME 0120-229/2018/12
Record Dates: First submitted 2020-09-24; First posted 2020-10-01 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Out-Of-Hospital Cardiac Arrest; lactic acid; Cardiopulmonary resuscitation; Survival
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: capillary lactate measurements — In this study capillary lactate will be measured every 10 minute during CPR.

SUMMARY:
Serial capillary lactate measurements during cardiopulmonary resuscitation (CPR) in patients with out-of-hospital cardiac arrest (OHCA).

DETAILED DESCRIPTION:
Capillary lactate measurements will be measured every ten minutes during CPR in OHCA.

ELIGIBILITY:
Inclusion Criteria:

* adults with OHCA

Exclusion Criteria:

* children with OHCA
* trauma
* hypothermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study will be eligible all patients with OHCA due to primary or secondary cardiac arrest.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
ROSC | 2 years
  In patients with ROSC the capillary lactate level will be lower compare to the non ROSC group.
Comparison between primary and secondary cardiac arrest | 2 years
  Initial and serial values of capillary lactate will be lower in patients with primary out-of- hospital cardiac arrest (OHCA)
No ROSC | 2 years
  Serial values of capillary lactate will be higher in patients without ROSC

CONTACTS AND LOCATIONS:
Overall Officials: Matej Strnad, MD, PhD, Study Director — University medical center Maribor
Locations (1):
- Community health center Maribor, Prehospital unit, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lurie KG, Nemergut EC, Yannopoulos D, Sweeney M. The Physiology of Cardiopulmonary Resuscitation. Anesth Analg. 2016 Mar;122(3):767-783. doi: 10.1213/ANE.0000000000000926. PMID 26562060
- [Background] Patil KD, Halperin HR, Becker LB. Cardiac arrest: resuscitation and reperfusion. Circ Res. 2015 Jun 5;116(12):2041-9. doi: 10.1161/CIRCRESAHA.116.304495. PMID 26044255
- [Background] Corral Torres E, Hernandez-Tejedor A, Suarez Bustamante R, de Elias Hernandez R, Casado Florez I, San Juan Linares A. Prognostic value of venous blood analysis at the start of CPR in non-traumatic out-of-hospital cardiac arrest: association with ROSC and the neurological outcome. Crit Care. 2020 Feb 22;24(1):60. doi: 10.1186/s13054-020-2762-5. PMID 32087761
- [Background] Sariaydin T, Corbacioglu SK, Cevik Y, Emektar E. Effect of initial lactate level on short-term survival in patients with out-of-hospital cardiac arrest. Turk J Emerg Med. 2017 May 15;17(4):123-127. doi: 10.1016/j.tjem.2017.05.003. eCollection 2017 Dec. PMID 29464213